CLINICAL TRIAL: NCT05509621
Title: The Effect of Positions on Physiological Parameters of Preterm Neonates Receiving Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Dilek Konukbay, Assistant professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-KONUKBAY-001
Record Dates: First submitted 2022-05-30; First posted 2022-08-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Preterm; Nursing Caries
Keywords: preterm neonate; position; mechanical ventilation; physiological parameters; nursing caries
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Preterm neonates to be included in the study will be placed in 5 different positions using a crossover design.In order not to repeat the order of positions,5 groups will be created as follows:ABCDE;BCDEA;CDEAB;DEABC;EABCD.The number of the groups created for not repeating the order of positions will be determined using the lottery method;Group1=CDEAB;Group2=BCDEA;Group3=EABCD;Group4=DEABC;Group5=ABCDE.Then,which position corresponds to which letter will be determined using the lottery method;A=quarter prone position,B=prone position,C=supine position,D=left lateral position,E=right lateral position.Afterward,40 preterm neonates will be randomly assigned to 5 groups using the block randomization method in line with the sample calculation. The order of the positions for the preterm neonate will be determined according to the position order of the group including the preterm infant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Supine position (Experimental): To determine the effect of supine position used during daily routine care in the neonatal intensive care unit on physiological parameters (oxygen saturation, heart rate, respiratory rate).
  Interventions: Other: The Effect of Supine Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns
- Prone position (Experimental): To determine the effect of prone position used during daily routine care in the neonatal intensive care unit on physiological parameters (oxygen saturation, heart rate, respiratory rate).
  Interventions: Other: The Effect of Prone Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns
- Left lateral position (Experimental): To determine the effect of left lateral position used during daily routine care in the neonatal intensive care unit on physiological parameters (oxygen saturation, heart rate, respiratory rate).
  Interventions: Other: The Effect of left lateral Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns
- Right lateral position (Experimental): To determine the effect of right lateral position used during daily routine care in the neonatal intensive care unit on physiological parameters (oxygen saturation, heart rate, respiratory rate).
  Interventions: Other: The Effect of right lateral Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns
- Quarter prone position (Experimental): To determine the effect of quarter prone position used during daily routine care in the neonatal intensive care unit on physiological parameters (oxygen saturation, heart rate, respiratory rate).
  Interventions: Other: The Effect of Quarter prone Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns

INTERVENTIONS:
Other: The Effect of Supine Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns — Preterm neonates who receive mechanical ventilation support and meet the study criteria will be provided with daily routine nursing care. Afterward, when it is time for positioning, the infant will be randomly placed in positions assigned according to the randomization. After positioning, data will not be collected for the first 30 minutes of each positioning in order to ensure the stability of the neonate. Starting from the 30th minute, the heart rate and oxygen saturation of the preterm neonate will be checked on the monitor at 15-minute intervals over the course of 90 minutes, and the respiratory rate will be counted and recorded for 1 minute by the researcher. For each position, the procedures will be repeated in the same way and the values will be recorded.
  Arms: Supine position
Other: The Effect of Prone Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns — Preterm neonates who receive mechanical ventilation support and meet the study criteria will be provided with daily routine nursing care. Afterward, when it is time for positioning, the infant will be randomly placed in positions assigned according to the randomization. After positioning, data will not be collected for the first 30 minutes of each positioning in order to ensure the stability of the neonate. Starting from the 30th minute, the heart rate and oxygen saturation of the preterm neonate will be checked on the monitor at 15-minute intervals over the course of 90 minutes, and the respiratory rate will be counted and recorded for 1 minute by the researcher. For each position, the procedures will be repeated in the same way and the values will be recorded.
  Arms: Prone position
Other: The Effect of left lateral Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns — Preterm neonates who receive mechanical ventilation support and meet the study criteria will be provided with daily routine nursing care. Afterward, when it is time for positioning, the infant will be randomly placed in positions assigned according to the randomization. After positioning, data will not be collected for the first 30 minutes of each positioning in order to ensure the stability of the neonate. Starting from the 30th minute, the heart rate and oxygen saturation of the preterm neonate will be checked on the monitor at 15-minute intervals over the course of 90 minutes, and the respiratory rate will be counted and recorded for 1 minute by the researcher. For each position, the procedures will be repeated in the same way and the values will be recorded.
  Arms: Left lateral position
Other: The Effect of right lateral Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns — Preterm neonates who receive mechanical ventilation support and meet the study criteria will be provided with daily routine nursing care. Afterward, when it is time for positioning, the infant will be randomly placed in positions assigned according to the randomization. After positioning, data will not be collected for the first 30 minutes of each positioning in order to ensure the stability of the neonate. Starting from the 30th minute, the heart rate and oxygen saturation of the preterm neonate will be checked on the monitor at 15-minute intervals over the course of 90 minutes, and the respiratory rate will be counted and recorded for 1 minute by the researcher. For each position, the procedures will be repeated in the same way and the values will be recorded.
  Arms: Right lateral position
Other: The Effect of Quarter prone Position on Physiological Parameters in Mechanically Ventilated Preterm Newborns — Preterm neonates who receive mechanical ventilation support and meet the study criteria will be provided with daily routine nursing care. Afterward, when it is time for positioning, the infant will be randomly placed in positions assigned according to the randomization. After positioning, data will not be collected for the first 30 minutes of each positioning in order to ensure the stability of the neonate. Starting from the 30th minute, the heart rate and oxygen saturation of the preterm neonate will be checked on the monitor at 15-minute intervals over the course of 90 minutes, and the respiratory rate will be counted and recorded for 1 minute by the researcher. For each position, the procedures will be repeated in the same way and the values will be recorded.
  Arms: Quarter prone position

SUMMARY:
This study was planned as an experimental study with a randomized crossover design to determine the effect of supine, prone, right lateral, left lateral, and quarter prone positions used during daily routine care in the neonatal intensive care unit on physiological parameters (oxygen saturation, heart rate, respiratory rate) of preterm neonates receiving mechanical ventilation.

DETAILED DESCRIPTION:
Preterm neonates face various adaptation problems starting from their birth due to their underdeveloped organ systems. A significant portion of preterm neonates need advanced care due to respiratory system problems, especially due to insufficient adaptation of the respiratory systems to the extrauterine environment, and the majority of them require mechanical ventilation. For these reasons, it is a priority to restore the respiratory functions of preterm neonates. To ensure the functionality of body systems in the developmental care of neonates in this process, the method of neonatal positioning, which is one of the individualized supportive developmental care methods, is necessary. The primary goal of positioning in neonatal intensive care units is to reduce the effects of pain and environmental stimuli caused by interventions for treatment and care for neonates and to help them cope with stress by maintaining their posture. Developmental positioning practices aim to support neuromotor development and minimize pain by maintaining the comfortable position of the neonate surrounded by the midline. The positioning has been shown to significantly affect the respiratory systems of neonates and affect oxygenation and lung ventilation. Change of position is also crucial in physiological and neurodevelopmental aspects for neonates receiving mechanical ventilation. It is important to reposition neonates since they remain in the same position all the time, which may lead to the accumulation of secretions and the formation of pressure sores. Positioning is an important factor in the development of neonates; therefore, correct positioning is critical for the comfort of neonates in the short and long term. Giving and maintaining a suitable position for neonates is an important nursing intervention. With developmentally supportive positioning applications, infants are positioned in supine, prone, lateral (right/left) and quarter prone positions. Considering these positions one by one, the supine position, where nursing care can be provided more easily, increases the sensory-motor activities of the neonate and reduces the energy consumption resulting from the infant's activities. Neonatal intensive care units mostly place neonates in the prone position since it has a positive effect on breathing, sleep quality, and behavioral conditions. The prone position makes the newborn feel safer with the adjustments made in the extrauterine environment. The lateral (right/left) position is one of the positions reducing the extensor effects of gravity and supporting the midline orientation of the hands and feet along with the head, which can be preferred in cases where the prone position cannot be used. In the quarter-prone position, neonates are placed in a functional position similar to the prone position but with one side of the body slightly elevated to encourage the synchronous movement of the thoracic and abdominal respiratory muscles. It has been observed that the quarter prone position provides similar advantages as the prone position by increasing lung compliance, tidal volume, respiratory rhythm, and oxygenation during sleep. Preterm neonates are placed in these positions in daily routine care of neonatal intensive care units.

The review of the relevant literature reveals studies comparing different groups regarding the positioning of preterm neonates receiving mechanical ventilators in the neonatal intensive care unit. These studies have mainly focused on the effect of supine, prone, right lateral and left lateral positions in preterm neonates receiving mechanical ventilation.

There is no study collectively comparing supine, prone, right lateral, left lateral and quarter prone positions used during daily routine care of preterm neonates receiving mechanical ventilation, which was aimed in this study. In this context, it was considered that evaluating the effect of supine, prone, right lateral, left lateral and quarter prone positions routinely used in the neonatal intensive care unit on the physiological parameters of preterm neonates receiving mechanical ventilation (oxygen saturation, heart rate, respiratory rate) and determining which position is more effective for preterm infants will contribute to the literature and guide the care provided by neonatal nurses.

Place And Tıme Of The Study:

This study was planned to be conducted in the Neonatal Intensive Care Unit of the University of Health Sciences Etlik Zubeyde Hanim Gynecology Training and Research Hospital between June 2022 and June 2023 after obtaining the necessary institutional and ethical committee approvals.

Hypotheses Of The Study:

Hypothesis 0(H0): There is no difference between prone, supine, right lateral, left lateral and quarter prone positioning of preterm infants in terms of physiological parameters of the infant.

Hypothesis 1.1(H1.1): Supine positioning of preterm infants is more effective in physiological parameters than other positions.

Hypothesis 1.2(H1.2): Prone positioning of preterm infants is more effective in physiological parameters than other positions.

Hypothesis 1.3(H1.3): Left lateral positioning of preterm infants is more effective in physiological parameters than other positions.

Hypothesis 1.4(H1.4): Right lateral positioning of preterm infants is more effective in physiological parameters than other positions.

Hypothesis 1.5(H1.5): Quarter prone positioning of preterm infants is more effective in physiological parameters than other positions.

Unıverse And Sample Of The Study:

The universe of the study comprised preterm neonates receiving mechanical ventilation in the Neonatal Intensive Care Unit of the University of Health Sciences Etlik Zubeyde Hanim Gynecology Training and Research Hospital. Multi-group comparisons were planned in the analysis of the hypotheses of the study and the sample size calculated according to the statistical method to be used was taken as a basis.

Using "G."Power version 3.1.9.2" software, the sample size was calculated at a confidence level of 95%. As a result of the analysis, α=0.05, the standardized effect size was calculated from a similar study conducted in this field. The minimum sample size was estimated as 8 subjects for each group when the effect size was taken as 0.72 (high), with theoretical power of 0.80. As evaluations will be carried out in 5 groups in this study, the minimum sample size was found to be 40.

ELIGIBILITY:
INCLUSION CRITERIA

* A gestational age of 28-36 weeks ,
* Receiving mechanical ventilation (non-intubated),
* Volunteer consent of the parents of the preterm neonate to participate in the study.

EXCLUSION CRITERIA

* Receiving mechanical ventilation and being intubated,
* Having any congenital and genetic disorders,
* Having a health problem that prevents positioning,
* Having a chest tube, umbilical catheter or PICC line,
* Receiving continuous sedative therapy, anticonvulsive therapy and cardiac drug therapy,
* Frequent changes in mechanical ventilator settings,
* A feeding frequency of more than three hours.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 1 year
  Beats per minute will be obtained using an electrocardiographic bedside monitor. An electrocardiographic bedside monitor will be placed on each of the babies.
Oxygen Saturation | 1 year
  Oxygen saturation (SpO2) will be obtained using an electrocardiographic bedside monitor. A separate electrocardiographic bedside monitor will be placed for each of the babies.
Respiratory Rate | 1 year
  Respiratory rate will be counted and recorded for 1 minute by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK KONUKBAY, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- University of Health Sciences Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Montgomery K, Choy NL, Steele M, Hough J. The effectiveness of quarter turn from prone in maintaining respiratory function in premature infants. J Paediatr Child Health. 2014 Dec;50(12):972-7. doi: 10.1111/jpc.12689. Epub 2014 Jul 13. PMID 25039401
- [Result] Utario Y, Rustina Y, Waluyanti FT. The Quarter Prone Position Increases Oxygen Saturation in Premature Infants Using Continuous Positive Airway Pressure. Compr Child Adolesc Nurs. 2017;40(sup1):95-101. doi: 10.1080/24694193.2017.1386976. PMID 29166184
- [Result] Yin T, Yuh YS, Liaw JJ, Chen YY, Wang KW. Semi-Prone Position Can Influence Variability in Respiratory Rate of Premature Infants Using Nasal CPAP. J Pediatr Nurs. 2016 Mar-Apr;31(2):e167-74. doi: 10.1016/j.pedn.2015.10.014. Epub 2015 Nov 21. PMID 26614613
- [Result] Brunherotti MA, Martinez EZ, Martinez FE. Effect of body position on preterm newborns receiving continuous positive airway pressure. Acta Paediatr. 2014 Mar;103(3):e101-5. doi: 10.1111/apa.12504. Epub 2013 Dec 20. PMID 24354904
- [Result] Gouna G, Rakza T, Kuissi E, Pennaforte T, Mur S, Storme L. Positioning effects on lung function and breathing pattern in premature newborns. J Pediatr. 2013 Jun;162(6):1133-7, 1137.e1. doi: 10.1016/j.jpeds.2012.11.036. Epub 2013 Jan 11. PMID 23312684
- [Result] Cakici M, Mutlu B. Effect of Body Position on Cardiorespiratory Stabilization and Comfort in Preterm Infants on Continuous Positive Airway Pressure. J Pediatr Nurs. 2020 Sep-Oct;54:e1-e8. doi: 10.1016/j.pedn.2020.06.015. Epub 2020 Jul 15. PMID 32680615